CLINICAL TRIAL: NCT01918449
Title: Follow-up of Patients With the Apnea-hypopnea Syndrome in Primary Care and Sleep Disorders Units. Equivalence Randomized Comparative Study on Compliance and Clinical Response.
Brief Title: Follow-up of Patients With Obstructive Sleep Apnea in Primary Care.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Fundacio Catalana de Pneumologia (Other)
Responsible Party: Principal Investigator, Ferran Barbe, MD, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI12/01499
Record Dates: First submitted 2013-07-23; First posted 2013-08-07 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: OSA
Keywords: OSA; CPAP treatment; primary care; efficacy
MeSH Terms: interventions — Primary Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep Unit group (No Intervention): This group will have standard follow up in sleep unit at 1, 3 and 6 month. These patients will also be instructed in hygienic-dietary measures, standard care of cardiovascular risk factors and sleep hygiene counseling.
- Primary Care group (Experimental): This group will have standard follow up in primary care at 1, 3 and 6 month. These patients will also be instructed in hygienic-dietary measures, standard care of cardiovascular risk factors and sleep hygiene counseling.
  Interventions: Other: Clinical follow up by general practitioners in primary care

INTERVENTIONS:
Other: Clinical follow up by general practitioners in primary care — The study evaluates two different setting to follow up patients with obstructive sleep apnea on CPAP treatment
  Arms: Primary Care group

SUMMARY:
The objective of the study is to compare the results of a coordinated and interactive program for the treatment, monitoring and control of patients with a moderate-severe diagnosis of Obstructive Sleep Apnea (OSA) and treated with positive continuous pressure (CPAP), with the currently established situation.

Methodology: Equivalence randomized comparative study . It will include patients with diagnosis of moderate-severe OSA (apnea-hypopnea Index >=15) that should start treatment with (CPAP). Participating center is Hospital Santa María-Arnau de Vilanova in Lleida (Spain).These patients will be randomized to two monitoring groups (1: monitoring in the Sleep disorders unit, 2: monitoring in primary care consultations) once the OSAS diagnosis has been made and it was indicated that treatment with CPAP. Patients Will be carried out in both groups the same follow-up visits in two study arms: basal, 1 month, 3 months and 6 months. Primary outcomes: number of hours of use per day (according to the accountant of the CPAP), so that use >= 4h/day is defined as good adherence to the treatment. Secondary outcomes: daytime sleepiness, patient satisfaction, Adverse events related to CPAP treatment. It will be collected demographic ,clinics and anthropometric variables. At the end of follow-up primary and secondary outcomes will be compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years old.
* Patients with OSA diagnosis performed in the sleep units
* Written informed consent signed.

Exclusion Criteria:

* Previous CPAP treatment for OSA diagnosis
* Psycho-physical inability to complete questionnaires.
* Presence of any previously diagnosed sleep disorders: narcolepsy, insomnia, chronic sleep deprivation, regular use of hypnotic or sedative medications and restless leg syndrome
* Patients with respiratory diseases (overlap syndrome, hypoventilation, restrictive diseases)
* A medical history that may interfere with the study objectives or, in the opinion of the investigator, compromise the conclusions.
* Any medical factor, social or geographical, that may jeopardize patient compliance.(e.g., alcohol consumption (more 80 gr/day in men and more than 60 gr / day in women), no fixed address, disorientation, or a history of non-compliance).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of hours of use per day of CPAP | Six month
  Number of hours of use per day of CPAP according to the internal clock of the CPAP device

SECONDARY OUTCOMES:
Daytime sleepiness | At baseline and at 6 month of follow-up
  Epworth Sleepiness Scale (ESS)
Patient satisfaction | Six month
  visual analog scale (0-10)
Adverse events | Six month
  Adverse events related to CPAP treatment
Quality of life | Baseline and at 6 month of follow up
  EuroQol
Cost-efficacy evaluation | Six month
  Qualys
Comorbidity index | Six month
  Charlson index
Blood pressure | Sixt month
  Office blood pressure
Lost of follow up | Six month
  Percentage of patients lost during follow up

OTHER OUTCOMES:
Body mass index | Six month

CONTACTS AND LOCATIONS:
Overall Officials: Ferran Barbe, MD, Study Director — Hospital Anrnau Vilanova- Santa Maria, Lleida (Spain); Cristina Esquinas, RN, MPH, Principal Investigator — Hospital Arnau Vilanova-Santa Maria, Lleida (Spain); Nuria Nadal, MD, Principal Investigator — Primary Care. National Health Institute. Lleida (Spain)
Locations (1):
- Hospital santa Maria, Lleida, Catalonia, Spain

REFERENCES:
- [Derived] Sanchez-de-la-Torre M, Nadal N, Cortijo A, Masa JF, Duran-Cantolla J, Valls J, Serra S, Sanchez-de-la-Torre A, Gracia M, Ferrer F, Lorente I, Urgeles MC, Alonso T, Fuentes A, Armengol F, Lumbierres M, Vazquez-Polo FJ, Barbe F; Respiratory Medicine Research Group. Role of primary care in the follow-up of patients with obstructive sleep apnoea undergoing CPAP treatment: a randomised controlled trial. Thorax. 2015 Apr;70(4):346-52. doi: 10.1136/thoraxjnl-2014-206287. PMID 25766689